CLINICAL TRIAL: NCT00596466
Title: An Open-Label Multicenter Extension Study To Determine Long Term Safety And Efficacy Of Pregabalin (Lyrica) As Monotherapy In Patients With Partial Seizures
Brief Title: Extension Study Of Long-Term Safety And Efficacy Of Pregabalin As Monotherapy (Lyrica) In Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081160
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-08

CONDITIONS: Epilepsy
Keywords: open-label; extension study; pregabalin; partial epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — pregabalin

SUMMARY:
This study will evaluate the long term safety and efficacy of pregabalin (Lyrica) when administered by itself (without any other anti-epileptic medication) to epilepsy patients for the treatment of partial seizures. This is an extension study to a previous clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Completed the previous protocol and wish to continue to receive pregabalin.
* Diagnosis of epilepsy with partial seizures

Exclusion Criteria:

* Early withdrawal from the previous protocol, an episode of status epliepticus, or primary generalized epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (32):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Suwanee, Georgia
  - Pfizer Investigational Site, Danville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Bowling Green, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Houma, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Pikesville, Maryland
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Great Falls, Montana
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Czechia (3):
  - Pfizer Investigational Site, Beroun
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Litomyšl
- Pfizer Investigational Site, New Territories, Hong Kong
- Ukraine (4):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Luhansk
  - Pfizer Investigational Site, Odesa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were eligible for the current study A0081160 (NCT00596466) if they adequately responded to pregabalin treatment in protocol A0081047 (NCT00524030).
Groups:
- Pregabalin: Pregabalin capsules, 300 milligrams per day (mg/day) twice daily (BID) for 24 weeks. Dose adjustments of pregabalin permitted (range of 150-600 mg, BID) based on investigator judgment.
Period: Overall Study
Arm/Group | Pregabalin
Started | 75
Enrolled, Treated | 73
Completed | 58
Not Completed | 17
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2
Not completed — Unpecified | 2
Not completed — Enrolled, not treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 75
Age, Customized [Number; unit: Participants]
  18-44 years | 48
  45-64 years | 23
  Greater than or equal to (≥) 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency
Time Frame: Baseline up to Week 28
Population: Not analyzed; Per protocol, seizure frequency data for individual participants were collected and reviewed but no statistical inferences were conducted because there was no comparator agent for this study.
Arm/Group | Pregabalin
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With (All Causality) Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to Week 28
Population: Safety analysis set population: all participants who received at least 1 dose of pregabalin.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 73
Participants
  Non-serious AEs | 30
  Serious AEs (SAEs) | 3

3. Primary Outcome: Number of Participants With Laboratory Test Values of Potential Clinical Importance
Description: Pre-defined criteria were established for each laboratory test (hematology, blood chemistry and urinalysis) to define the values that would be identified as of potential clinical importance.
Time Frame: Baseline up to Week 28
Population: Safety analysis set population; Number of participants analyzed (N): participants with at least one observation of any given laboratory test while on study.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 72
Participants | 17

ADVERSE EVENTS:
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 3/73
Other Adverse Events (participants affected / at risk) | 14/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=73)
Road traffic accident (Injury, poisoning and procedural complications) | 1
Convulsion (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=73)
Nausea (Gastrointestinal disorders) | 4
Weight increased (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Convulsion (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.